CLINICAL TRIAL: NCT07124702
Title: Cessation of Dual Use of Cigarettes and E-cigarettes During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Xiaozhong Wen, Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00008644; UL1TR001412 (NIH)
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Dual Use of Cigarettes and E-cigarettes; Gestational Weight Gain; Birth-weight-for-gestational-age z Score
Keywords: Randomized Controlled Trial; Tobacco use; Electronic cigarette; Pregnancy; Intervention
MeSH Terms: conditions — Vaping; Gestational Weight Gain; Tobacco Use

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simultaneous cessation intervention (Experimental): This simultaneous cessation intervention group will target CCs and ECs at the same time. Participants in this group will receive a multi-component cessation intervention, including behavior counseling, biomarker feedback via monitoring changes in levels of exposure to nicotine (urine cotinine) and CC smoke (breath carbon monoxide), and contingent financial incentives for biochemically verified abstinence.
  Interventions: Behavioral: Simultaneous cessation intervention
- Stepwise cessation intervention (Experimental): This stepwise cessation intervention group will first target CCs and then target ECs after quitting CCs. Participants in this group will receive a multi-component cessation intervention, including behavior counseling, biomarker feedback via monitoring changes in levels of exposure to nicotine (urine cotinine) and CC smoke (breath carbon monoxide), and contingent financial incentives for biochemically verified abstinence.
  Interventions: Behavioral: Stepwise cessation intervention
- Control group (Active Comparator): Participants assigned to the control group will receive behavior counseling only. They will complete the same number of study visits as their counterparts in the intervention groups.
  Interventions: Behavioral: Behavior counseling only

INTERVENTIONS:
Behavioral: Simultaneous cessation intervention — This simultaneous cessation intervention group will target CCs and ECs at the same time. Participants in this group will receive a multi-component cessation intervention, including behavior counseling, biomarker feedback via monitoring changes in levels of exposure to nicotine (urine cotinine) and CC smoke (breath carbon monoxide), and contingent financial incentives for biochemically verified abstinence.
  Arms: Simultaneous cessation intervention
Behavioral: Stepwise cessation intervention — This stepwise cessation intervention group will first target CCs and then target ECs after quitting CCs. Participants in this group will receive a multi-component cessation intervention, including behavior counseling, biomarker feedback via monitoring changes in levels of exposure to nicotine (urine cotinine) and CC smoke (breath carbon monoxide), and contingent financial incentives for biochemically verified abstinence.
  Arms: Stepwise cessation intervention
Behavioral: Behavior counseling only — Participants assigned to the control group will receive behavior counseling only. They will complete the same number of study visits as their counterparts in the intervention groups.
  Arms: Control group

SUMMARY:
We propose a randomized controlled trial to develop and evaluate a cessation program with two different strategies for dual users during pregnancy. We plan to enroll 45 pregnant mothers (≤20 gestational weeks) with low household incomes from the Western NY region. To be eligible, they must be currently dual using CCs and nicotine-containing ECs. These mothers will be randomized into one of three groups: 1) simultaneous cessation intervention group (N=15), 2) stepwise cessation intervention group (N=15), and 3) control group (N=15). We hypothesize that nicotine abstinence rates at 8 weeks after randomization will be higher in the intervention groups than in the control group.

DETAILED DESCRIPTION:
Study overview. We propose a pilot randomized controlled trial (RCT) to develop and test a cessation program for dual users during pregnancy. We will enroll 45 Western New York pregnant mothers (≤20 weeks gestational age) with low household incomes who are currently dual-using CCs and nicotine-containing ECs. These mothers will be randomized into one of three groups: 1) simultaneous cessation intervention (N=15), 2) stepwise cessation intervention (N=15), and 3) control group (N=15). Both intervention groups will receive a multi-component intervention, including behavior counseling, biomarker feedback, and contingent financial incentives for biochemically verified abstinence. However, the two intervention groups will have different orders of cessation targets: the simultaneous cessation group will target CCs and ECs at the same time, whereas the stepwise cessation group will first target CCs and then target ECs after quitting CCs. The control group will only receive behavior counseling. Mothers will be followed throughout pregnancy until delivery. The primary outcome is nicotine abstinence at 8 weeks after randomization.

Randomization. After the pre-test visit, participants who are still dual using CCs and ECs will be randomized into one of three groups: 1) simultaneous cessation intervention group, 2) stepwise cessation intervention group, and 3) control group. A computer will be used to generate balanced-permuted blocks with a block size of 9 and a 3-3-3 ratio, which can ensure equal numbers of participants across the three groups throughout the project. The study biostatistician will create the sequences a priori and then apply them using a workflow and database software system.

Sample size. Based on the literature and our previous intervention, we estimate the dual-use nicotine abstinence rate at 8 weeks after randomization (the primary maternal outcome) to be 30% in the intervention groups versus 10% in the control group. Accordingly, we need 62 participants per group to detect a significant difference in nicotine abstinence with 80% power at a significance level of 0.05 (Aim 1). Therefore, 15 participants per group for this pilot study should provide a sufficient sample size to test study feasibility, recruitment, and retention and yield preliminary data on intervention efficacy and the magnitude of group differences in health outcomes to support an NIH R01 grant application for a large project.

Statistical analysis. We will first conduct descriptive analyses to determine if transformations are necessary, and then run bivariate analyses. We will compare the distributions of covariates above across the 3 randomized groups. Only the unbalanced covariates that predict smoking/vaping abstinence will be controlled in data analyses. We will use Intention-to-Treat analysis, i.e., including all women as assigned at randomization. Multiple imputations with 20 replicates will be used to impute missing data on outcomes or covariates.36 Sensitivity analysis will be conducted by conservatively assuming participants lost in the follow-up to be current dual users.

We will use Chi-square tests to compare categorical outcomes (e.g., maternal nicotine abstinence rates) and analysis of variance to compare continuous outcomes (e.g., infant birth-weight-for-gestational-age z-score) across groups. Then, we will use multivariable logistic and linear regression models to fit categorical and continuous outcomes, respectively. A propensity score approach will be used to control confounders, including socio-demographics, pregnancy-related characteristics, and other substance use. The model will include group assignment (simultaneous cessation intervention vs. control, stepwise cessation intervention vs. control, or simultaneous vs. stepwise cessation intervention), fidelity of intervention delivery, adherence to intervention, and a propensity score derived from all unbalanced covariates. We will estimate the group differences in nicotine abstinence rates and odds ratios from the regression model.

ELIGIBILITY:
Inclusion Criteria:

* Less than 21 weeks pregnant to ensure adequate time for intervention;
* 18 years or older;
* Actively using both cigarettes and electronic cigarettes (e-cigarettes);
* Willing to receive cessation information;
* Able to read, understand, and speak English;
* Having a low household income defined as ≤185% of the federal poverty level.

Exclusion Criteria:

* Teen pregnancy (<18 y);
* Unstable housing;
* Uncontrolled mental health disorders;
* Non-English speakers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Nicotine abstinence | 8 weeks after randomization, at the end of pregnancy
  Research staff who are blinded to the participant's group assignment will administer a timeline follow-back interview (trained by the PI, Dr. Wen) to assess the participant's recent smoking and vaping history. Based on self-reports, we will classify smoking and vaping status in the past 7 days (7-day point prevalence) prior to the outcome assessment visits at pre-test, 8 weeks after randomization, and at the end of pregnancy. To confirm self-reported complete nicotine abstinence (i.e., abstinence from both ECs and CCs), 5.0 mL of urine samples will be collected at study visits in the 8th week after randomization and at the end of pregnancy (approximately 35 weeks). An HPLC-MS/MS assay will be used as a gold standard test to determine urine cotinine levels.

SECONDARY OUTCOMES:
The time needed to achieve nicotine abstinence | 8 weeks after randomization, at the end of pregnancy
  We define the time needed to achieve nicotine abstinence as the interval between the day of randomization and the first day of complete nicotine abstinence ("not even a puff") without any relapse until birth delivery.
The mother's gestational weight gain | Right before delivery
  Total gestational weight gain (GWG) will be calculated as the difference between weight right before delivery and pre-pregnancy weight. Based on 2009 the Institute of Medicine (IOM) guidelines, we will define inadequate GWG as total GWG less than 28, 25, 15, and 11 pounds for underweight (pre-pregnancy BMI<18.5 kg/ m2), normal weight (BMI 18.5-24.9), overweight (BMI 25-29.9), and obese mothers (BMI ≥30), respectively.
The infant's birth-weight-forgestational- age z score | At birth
  We will obtain the infant's gestational age, clinical measures on weight, length, and head circumference at birth from delivery records. Gestational age will be calculated as the interval between the self-reported last menstrual period and delivery date. We will calculate the infant's birth-weight-for-gestational-age z score and percentile for the same sex and gestational age. SGA will be defined as birth weight below the 10th percentile.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Wen, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Confidentiality reasons.